CLINICAL TRIAL: NCT07054476
Title: The Effects of Intermittent and Continuous Enteral Nutrition on Glycaemic Control andSome Metabolic Parameters in Adult Critical Patients With Diabetes Receiving Clinical Nutritional Therapy
Brief Title: Intermittent vs Continuous Enteral Nutrition in Glycaemic Control of Diabetic ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Irem Nur Aksoylu, Dietitian, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-93471371-514.99-221892499
Record Dates: First submitted 2025-05-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Glycemic Control for Diabetes Mellitus; Glycaemia
Keywords: Intensive care; continuous enteral nutrition; intermittent enteral nutrition; diabetes; metabolic parameters
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model in which participants were randomized into two separate intervention groups: Continuous Enteral Nutrition (CE) and Intermittent Enteral Nutrition (IE). Each participant remained in their assigned group for the entire 7-day intervention period without crossover between groups.
Who Masked: Participant
Masking Description: Participants were blinded to group assignment. Neither the continuous (CE) nor intermittent (IE) feeding method was disclosed to the patients due to their critical illness status. However, care providers, investigators, and outcome assessors were aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Enteral Nutrition Group (CE) (Active Comparator): Participants in this arm received continuous enteral nutrition based on the existing hospital protocol. After reaching 80% of the target energy requirements without signs of feeding intolerance, patients were provided with diabetic-specific enteral formula administered continuously. Energy needs were calculated using the ESPEN guideline (25 kcal/kg/day).
  Interventions: Other: Continuous Enteral Nutrition (CE)
- Intermittent Enteral Nutrition (IE) (Experimental): Participants in this arm received intermittent enteral nutrition as part of the study protocol. After reaching 80% of the target energy requirements without signs of feeding intolerance, patients were provided with diabetic-specific enteral formula administered in 5 discrete sessions across the 24-hour period, with scheduled breaks between feeding sessions. Energy needs were calculated using the ESPEN guideline (25 kcal/kg/day). This intervention was designed to compare the effects of intermittent feeding schedules against continuous feeding in critically ill diabetic patients.
  Interventions: Other: Intermittent Enteral Nutrition

INTERVENTIONS:
Other: Intermittent Enteral Nutrition — Intermittent Enteral Nutrition (IE):
  The intervention involves intermittent enteral nutrition using a diabetic-specific enteral formula, administered in 5 separate sessions daily with scheduled breaks between feedings. Each feeding session is followed by a break (1-2 hours). Energy needs are calculated based on the ESPEN guideline (25 kcal/kg/day). This protocol is designed to assess the effects of intermittent feeding in critically ill diabetic patients.
  Arms: Intermittent Enteral Nutrition (IE)
Other: Continuous Enteral Nutrition (CE) — Continuous Enteral Nutrition (CE): The intervention involves continuous enteral nutrition provided via a diabetic-specific enteral formula, administered 24 hours a day with 1-hour breaks between feeding sessions. The feeding rate starts at 40cc per hour and is gradually increased based on tolerance. Energy needs are calculated using the ESPEN guideline (25 kcal/kg/day).
  Arms: Continuous Enteral Nutrition Group (CE)

SUMMARY:
The goal of this clinical trial is to learn if intermittent or continuous enteral nutrition applications can improve glycemic control and affect certain metabolic parameters in adult critically ill patients with diabetes receiving clinical nutrition therapy. The main questions it aims to answer are:

Does intermittent enteral nutrition lead to better glycemic control compared to continuous enteral nutrition?

How do intermittent and continuous enteral nutrition applications affect metabolic parameters such as serum insulin levels, lipid profile, and inflammatory markers?

Researchers will compare intermittent and continuous enteral nutrition groups to see if one method is more effective in improving glycemic control and metabolic outcomes.

Participants will:

Receive either intermittent or continuous enteral nutrition as part of their clinical nutrition therapy

Have regular blood tests to monitor blood glucose, insulin, lipid profile, and inflammatory markers

Be monitored for glycemic variability and metabolic changes during their ICU stay

DETAILED DESCRIPTION:
This randomized controlled clinical trial was conducted in the 25-bed tertiary intensive care unit of the Anesthesiology and Reanimation Department at Ankara Training and Research Hospital. Ethical approval was obtained from the institutional review board, and written informed consent was provided by the legal representatives of all participants. The study was carried out between December 2023 and June 2024, including 25 adult diabetic patients (14 males, 11 females; mean age: 73.44 ± 8.97 years) who were receiving clinical nutrition therapy in the ICU.

The purpose of this study was to compare the effects of continuous enteral nutrition (CE) and intermittent enteral nutrition (IE) on glycemic control and selected metabolic parameters. Sample size was calculated using G*Power software, indicating that a minimum of 24 participants (12 per group) would be needed to detect a large effect size (1.39) with 80% power and a 5% type I error rate.

All patients initially began enteral feeding at 40 mL/hour according to standard ICU protocol, with gradual increases based on individual tolerance. Once patients reached 80% of their estimated energy requirement without feeding intolerance, they were randomized into one of two groups:

CE group (Control, n=12): Received enteral nutrition in a near-continuous fashion with scheduled breaks.

IE group (n=13): Received nutrition in defined intermittent periods, alternating with fasting intervals.

Energy needs were estimated using the ESPEN guideline formula (25 kcal/kg/day), and a diabetic-specific enteral formula was administered accordingly.

Blood glucose levels were measured five times per day (06:00, 11:00, 16:00, 21:00, and 01:00) using a bedside glucometer. In addition, all participants had the following data collected:

Clinical scores: SOFA, mNUTRIC, and APACHE II

Baseline and Day 7 measurements of serum total cholesterol and triglycerides

Daily laboratory parameters: serum glucose, ALT, AST, GGT, albumin, CRP, BUN, creatinine, sodium, and potassium

The intervention lasted for 7 days and aimed to evaluate whether the method of enteral nutrition delivery (CE vs. IE) affects metabolic responses and glycemic outcomes in diabetic ICU patients. Findings from this study may help inform nutritional strategies in critical care for individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older

Diagnosis of diabetes

Receiving enteral nutrition

Indication for at least 7 days of ICU admission to perform the study

Exclusion Criteria:

* Under 18 years old

Having specific needs that would require a completely different type of treatment, such as cancer or cystic fibrosis

Pregnancy

Expected to stay in the ICU for less than 7 days

Receiving oral feeding or TPN (Total Parenteral Nutrition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Levels (mg/dL) | Five measurements per day at 06:00, 11:00, 16:00, 21:00, and 01:00, for 7 consecutive days
  The primary outcome measure will be the effect of continuous versus intermittent enteral nutrition on glycemic control in critically ill diabetic patients. Blood glucose levels will be monitored 5 times per day using a glucose meter (GlucoNavii, Korea). Measurements will be taken at the following times: 06:00, 11:00, 16:00, 21:00, and 01:00.

SECONDARY OUTCOMES:
Serum Triglyceride Levels (mg/dL) | Baseline (Day 1) and Day 7
  Serum triglyceride levels will be measured to assess the impact of enteral nutrition on lipid metabolism. Blood samples will be collected at baseline (Day 1) and on Day 7 of intervention.
Serum Cholesterol Levels (mg/dL) | Baseline (Day 1) and Day 7
  Serum cholesterol levels will be measured to assess the impact of enteral nutrition on lipid metabolism. Blood samples will be collected at baseline (Day 1) and on Day 7 of intervention.
Serum Albumin Levels (g/dL) | Daily measurements for 7 consecutive days
  Serum albumin levels will be assessed as an indicator of nutritional status and response to enteral feeding protocols. Blood samples will be drawn daily for 7 days.
Serum CRP (C-Reactive Protein) Levels (mg/L) | Daily measurements for 7 consecutive days
  Serum CRP levels will be monitored to evaluate the inflammatory response in critically ill patients receiving enteral nutrition. Blood samples will be drawn daily for 7 days.
Serum Alanine aminotransferase (ALT) Levels (U/L) | Daily measurements for 7 consecutive days
  Serum levels of ALT will be monitored to assess liver function and potential liver injury in response to enteral nutrition protocols. Blood samples will be drawn daily for 7 days.
Serum Aspartate aminotransferase (AST) Levels (U/L) | Daily measurements for 7 consecutive days
  Serum levels of AST will be monitored to assess liver function and potential liver injury in response to enteral nutrition protocols. Blood samples will be drawn daily for 7 days.
Serum Gamma glutamyl transferase (GGT) Levels (U/L) | Daily measurements for 7 consecutive days
  Serum levels of GGT will be monitored to assess liver function and potential liver injury in response to enteral nutrition protocols. Blood samples will be drawn daily for 7 days.
Serum Blood Urea Nitrogen (BUN) Levels (mg/dL) | Daily measurements for 7 consecutive days
  Serum levels of BUN will be assessed to evaluate kidney function in critically ill patients receiving enteral nutrition. Blood samples will be drawn daily for 7 days.
Serum Creatinine Levels (mg/dL) | Daily measurements for 7 consecutive days
  Serum levels of creatinine will be assessed to evaluate kidney function in critically ill patients receiving enteral nutrition. Blood samples will be drawn daily for 7 days.
Sequential Organ Failure Assessment (SOFA) Score | First day of admission to the ICU
  The SOFA score evaluates the function of six organ systems-respiratory, cardiovascular, hepatic, coagulation, renal, and neurological-in critically ill patients. It is used to monitor the extent of organ dysfunction and predict clinical outcomes in the intensive care unit (ICU). Unit of Measure: Score (0-24 scale) Interpretation: Higher scores indicate greater organ dysfunction and worse prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Akyol Mutlu, Prof., Study Director — Hacettepe University
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Although ethical approval was obtained for the study, the individual participant data (IPD) were not anonymized during data entry and were recorded in SPSS with identifiable information such as names and surnames. Therefore, due to concerns regarding participant confidentiality and data protection, there is no plan to share the IPD.

REFERENCES:
- [Background] Ren CJ, Yao B, Tuo M, Lin H, Wan XY, Pang XF. Comparison of sequential feeding and continuous feeding on the blood glucose of critically ill patients: a non-inferiority randomized controlled trial. Chin Med J (Engl). 2021 Jul 20;134(14):1695-1700. doi: 10.1097/CM9.0000000000001684. PMID 34397596